CLINICAL TRIAL: NCT04105790
Title: The Acceptability and Effectiveness of Stepped Care Psychoeducation Classes in Rural Manitoba
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Pamela Black, Assistant Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2019:311
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Depressive Symptoms; Anxiety Symptoms
Keywords: Stepped Model of Care; Class-Based Intervention
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The overarching design of the proposed study is a formative program evaluation using a case series methodology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants in class-based mental health intervention.
  Interventions: Behavioral: Cognitive Behavioural Therapy with Mindfulness classes

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy with Mindfulness classes — The standard CBTm protocol is comprised of four 90-minute classes offered virtually via videoconferencing once a week for four consecutive weeks. The classes cover topics including mindfulness, cognitive therapy principles, behaviour therapy principles, managing anger, assertiveness, problem solving, goal setting, and evidence-based self-help resources. They are lecture-based but also involve experiential elements, such as mindfulness activities and practice of cognitive therapy strategies. Participants are assigned daily homework between each class to practice the strategies taught in session.

SUMMARY:
This study will examine the acceptability and effectiveness of using a stepped care treatment model, and specifically, the CBTm classes, in a rural population. The introduction of CBTm classes, developed in Winnipeg and used in outpatient mental health clinics there, is new to Adult Community Mental Health in the Prairie Mountain Health region. This research is being done to explore whether this is a treatment model that is effective at reducing symptoms of anxiety and depression and also whether it affects the workload for Community Mental Health Workers in a more rural area. Further, this research is being done to explore whether clients perceive this form of services to be useful and acceptable.

DETAILED DESCRIPTION:
This study will evaluate the acceptability and effectiveness of class-based psychoeducation as the first step of a stepped care model in a community mental health program. In April of 2019, the Prairie Mountain Health (PMH) Adult Community Mental Health programs (both Northern and Southern regions) instituted a change to their existing service model. Previously, all individuals who sought access to public mental health services underwent an intake interview and were subsequently assigned a community mental health worker (CMHW) with whom they met for individual counselling. Due to the ever-increasing demand for services, CMHWs were required to manage large caseloads which resulted in extended periods between counselling appointments and strain on care providers. In an effort to introduce a stepped-care framework to mitigate workload, the Adult Community Mental Health programs in PMH North and South began to offer psychology-led psychoeducation classes as a step below individual counselling. Specifically, the Cognitive Behavioural Therapy with Mindfulness (CBTm) classes, developed at the University of Manitoba by Sareen, Sala, Wong, Whitney, and Kinley (2016), were delivered. This program is comprised of four 90-minute sessions that deliver information about basic cognitive and behavioural therapy principles and effective self-help resources. It was developed to offer services to clients on the waitlist for outpatient mental health services in Winnipeg and preliminary research on this program has demonstrated that it is an acceptable form of treatment and effectively reduces symptoms of anxiety and depression (with a small to medium effect).

As the change in the service delivery model and the introduction of large psychoeducation classes in PMH's Adult Community Mental Health programs is novel, evaluation of this change is warranted. This study will examine foundational program variables including retention, acceptability, and effectiveness (see Thakur, Bolton, & Sareen, 2018). Assessing these factors will provide critical information about the potential for further development of a stepped care model, including the CBTm program, in this rural health region and afford the opportunity to compare outcome measures in a rural setting to those from an urban centre (data published by Thakur et al., 2018). In order to further increase access to services, the program was also intended to be delivered to remote rural sites via telehealth; exploration of the acceptability and efficacy of telehealth use in service delivery also merits assessment. However, at the start of the COVID-19 pandemic, in-person and MBTelehealth CBTm classes were suspended to abide by provincial physical distancing guidelines. Moving forward, the CBTm classes will be offered via MS Teams, a virtual videoconferencing platform for all attendees, allowing individuals to participate via videoconference or telephone from their preferred location within Manitoba.

The research questions and hypotheses are as follows:

1. Is the implementation of CBTm as the first step in a stepped model acceptable to rural clients? The investigators hypothesize that class-based clinical service will be acceptable to rural clients as it will increase their access to valuable mental health services in their region; this will be demonstrated in a high rate of retention and positive feedback from participants.
2. How are issues unique to rural settings, such as concerns about confidentiality and virtual delivery of programming, in a class-based setting viewed by rural clients? The investigators anticipate initial concerns about confidentiality and virtual service delivery related to the nature of the rural setting.
3. Are class-based clinical services (i.e., CBTm) effective for reducing symptoms of depression and anxiety for participants living in rural areas? Consistent with previous research, the investigators anticipate a small to medium effect size in the decrease of symptoms of depression and anxiety and increased incorporation of cognitive behavioural strategies into daily life.

ELIGIBILITY:
Inclusion Criteria:

* Adult clients (18+ years) accessing community mental health services for symptoms of depression and anxiety, and
* Interest in attending Cognitive Behaviour Therapy with Mindfulness classes.

Exclusion Criteria:

* Active psychosis or mania,
* Acutely elevated suicide risk,
* Severe cognitive impairment, and/or
* Non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Change measure (baseline, week 2, week 3, and week 4)
  Self-report measure of severity of depressive symptoms to be completed prior to each intervention class. Each of the 9 items is scored 0-3 (0 = not at all; 3 = nearly every day), yielding a total between 0 and 27, with higher scores representing increased severity of depression symptoms.
Generalized Anxiety Disorder-7 (GAD-7) | Change measure (baseline, week 2, week 3, and week 4)
  Self-report measure of severity of generalized anxiety symptoms to be completed prior to each intervention class. Each of the 7 items is scored 0-3 (0 = not at all; 3 = nearly every day), yielding a total between 0 and 21, with higher scores representing increased severity of generalized anxiety symptoms.
Acceptability Survey | Change measure (baseline and week 4)
  Self-report measure of the acceptability of different elements of the intervention to be completed prior to the first and fourth classes.
Class Evaluation Form | Data collected weekly throughout the four weeks of study enrolment
  Self-report measure of the acceptability of different elements of the intervention to be completed prior to the first and fourth intervention classes.

SECONDARY OUTCOMES:
Clinical Global Impression scale (CGI) | Change measure (baseline at week 2, week 3, and week 4)
  Self-report measure of improvement in symptoms to be completed prior to intervention classes 2, 3 and 4. The single item is scored 1-7 (1 = very much improved; 7 = very much worse), yielding a total between 1 and 7, with higher scores representing a worsening of symptoms.
Cognitive Behaviour Therapy Skills Questionnaire (CBTSQ) | Change measure (baseline, week 2, week 3, and week 4)
  Self-report measure of the extent of participants' learning and implementation of cognitive and behavioural coping skills to be completed prior to each intervention class. Each of the 16 items is scored 1-5 (1 = I don't do this; 5 = I always do this). The measure is comprised of two subscales, (1) Behavioural Activation (7 questions) and (2) Cognitive Restructuring (9 questions); item scores are summed to yield subscale scores, with higher scores indicating increased implementation of the respective subscale skills. The two subscales can be summed to create a total score, yielding a total between 16 and 80, with higher scores representing increased implementation of both sets of skills.
Treatment Acceptability/Adherence Scale (TAAS) | Change measure (baseline, week 2, week 3, and week 4)
  Self-report measure related to perceptions of the therapy and participants' ability to engage in the skills taught during the class to be completed prior to intervention classes 2, 3, and 4. Each of the 10 items is scored from 1-7 (1 = disagree strongly; 7 = agree strongly), yielding a total between 10 and 70, with higher scores representing positive perceptions of treatment acceptability and adherence.
Homework Record | Data collected weekly throughout the four weeks of study enrolment
  Self-report measure of homework completion and skills practice to be completed prior to intervention classes 2, 3 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Black, PhD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Prairie Mountain Health South - Adult Community Mental Health, Brandon, Manitoba
  - Prairie Mountain Health North - Community Mental Health, Dauphin, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sareen, J., Sala, T., Wong, J., Whitney, D., & Kinley, J. (2016). CBTm facilitator training manual. Retrieved from http://cbtm.ca/wp-content/uploads/2017/08/Facilitators_binder.pdf
- [Background] Thakur VK, Wong JY, Randall JR, Bolton JM, Parikh SV, Mota N, Whitney D, Palay J, Kinley J, Diocee S, Sala T, Sareen J. An evaluation of large group cognitive behaviour therapy with mindfulness (CBTm) classes. BMC Psychiatry. 2019 May 3;19(1):132. doi: 10.1186/s12888-019-2124-5. PMID 31053070
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Jacob KL, Christopher MS, Neuhaus EC. Development and validation of the cognitive-behavioral therapy skills questionnaire. Behav Modif. 2011 Nov;35(6):595-618. doi: 10.1177/0145445511419254. Epub 2011 Sep 5. PMID 21893554
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Milosevic I, Levy HC, Alcolado GM, Radomsky AS. The Treatment Acceptability/Adherence Scale: Moving Beyond the Assessment of Treatment Effectiveness. Cogn Behav Ther. 2015;44(6):456-69. doi: 10.1080/16506073.2015.1053407. Epub 2015 Jun 19. PMID 26091250
- See also: Website for Cognitive Behavioural Therapy with Mindfulness classes — http://cbtm.ca